CLINICAL TRIAL: NCT06635135
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Study of Adjunctive Aticaprant Plus an Antidepressant for Relapse Prevention in Major Depressive Disorder (MDD) With Moderate-to-severe Anhedonia
Brief Title: A Study of Aticaprant Plus an Antidepressant to Prevent Return of Depression Symptoms in Participants With Major Depressive Disorder Who Experience a Loss of Interest and Pleasure
Acronym: VENTURA-5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early study termination due to insufficient efficacy.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67953964MDD3005; 67953964MDD3005 (Other: Janssen Research & Development, LLC); 2024-511057-22-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-09; First posted 2024-10-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorder, Major; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aticaprant (Experimental)
  Interventions: Drug: Aticaprant
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aticaprant — Aticaprant will be administered orally.
  Other Names: JNJ-67953964
  Arms: Aticaprant
Other: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess how well aticaprant works compared to placebo when given in addition to antidepressant therapy (selective serotonin reuptake inhibitor [SSRI] or serotonin-norepinephrine reuptake inhibitor [SNRI]) in preventing return of depression symptoms in participants with major depressive disorder who experience a loss of interest and pleasure and who achieve a stable response after treatment with adjunctive aticaprant.

ELIGIBILITY:
Inclusion Criteria:

* Be medically stable based on physical examination (including a brief neurologic examination), medical history, vital signs (including blood pressure), and 12-lead electrocardiogram (ECG) performed at screening and OL baseline
* Be medically stable based on clinical laboratory tests performed at screening
* Meet DSM-5 diagnostic criteria for recurrent or single episode MDD, without psychotic features upon clinical assessment and confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) Axis I Disorders-Clinical Trials version (SCID-CT)
* Have symptoms of anhedonia based on clinical assessment and confirmed by presence of anhedonia (positive response to major depressive episode (MDE) module symptom Item 2) on the SCID-CT at screening

Exclusion Criteria:

* Has had no response to 2 or more consecutive antidepressant treatments administered at adequate dose and duration in the current episode of depression including the current selective SSRI/SNRI assessed using the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH ATRQ)
* Has a history or evidence of clinically meaningful noncompliance with current antidepressant therapy
* Has a history of moderate-to-severe substance use disorder including alcohol use disorder according to DSM-5 criteria within 6 months before screening
* Has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 3 months prior to the start of the screening phase
* Has cognitive impairment per investigator judgment that would render the informed consent invalid or limit the ability of the participant to comply with the study requirements

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Time from Randomization into Double Blind (DB) Treatment Maintenance Phase to First Documentation of Relapse | From randomization in DB phase to first relapse during the DB maintenance phase (that is [i.e.], up to 2 years 2 months in DB phase)
  Time from randomization into the DB treatment maintenance phase to the first documentation of a depression relapse event will be reported.

SECONDARY OUTCOMES:
Change in Sexual Function (SF) Measured by Changes in Sexual Functioning Questionnaire - Short-Form (CSFQ-14) Total Score From DB Baseline to End of Week 4 of the DB Treatment Maintenance Phase | From Week 16 (DB baseline) to end of week 4 of DB treatment maintenance phase (i.e., up to Week 20 of the study)
  Change in SF measured by CSFQ-14 total score from DB baseline to end of week 4 of DB treatment maintenance phase will be reported.
Change from DB baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score to End of DB Treatment Maintenance Phase | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in the MADRS total score to end of DB treatment maintenance phase will be reported.
Percentage of Participants With Remission of Depressive Symptoms MADRS Total Score Less Than or Equal to (<=) 10 | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Percentage of participants with remission of depressive symptoms defined as MADRS total score <= 10 will be reported.
Percentage of Participants With Remission of Depressive Symptoms (PHQ-9 Total Score <=4) | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Percentage of participants with remission of depressive symptoms defined by Patient Health Questionnaire, 9-item (PHQ-9) total score <=4 will be reported.
Percentage of Participants With Response of Depressive Symptoms Based on MADRS Total Score Over Time | For open-label (OL) treatment phase: Baseline (Day 1) up to Week 16; For DB Phase: From Week 16 (DB Baseline) up to 2 years 2 months in DB phase
  Percentage of participants with response defined as greater than or equal to (>=) 50% improvement in the MADRS total score over time will be reported.
Percentage of Participants With Response of Depressive Symptoms Based on PHQ-9 Total Score Over Time | For OL treatment phase: Baseline (Day 1) up to Week 16; For DB Phase: From Week 16 (DB Baseline) up to 2 years 2 months in the DB phase
  Percentage of participants with response of depressive symptoms based on PHQ-9 total score over time will be reported.
Change from DB Baseline in the Clinical Global Impression - Severity (CGI-S) Depression Scale Score | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in the CGI-S depression scale score will be reported.
Change from DB Baseline in PHQ-9 Total Score | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in PHQ-9 total score will be reported.
Change From DB Baseline in Anhedonia as Assessed by the Dimensional Anhedonia Rating Scale (DARS) Total Score | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in Anhedonia as assessed by the DARS total score will be reported.
Change from DB Baseline in Snaith-Hamilton Pleasure Scale (SHAPS) Score to End of DB Treatment Phase | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in SHAPS score to end of DB treatment phase will be reported.
Percentage of Participants who Relapse and Have Evidence of Anhedonia Over Time | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Percentage of participants who relapse and have evidence of anhedonia over time will be reported.
Change from DB Baseline in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) Total Score Over Time | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in the GAD-7 total score over time will be reported.
Change from DB Baseline in SF Measured by CSFQ-14 Total Score and SF Domain Scores Over Time | From Week 16 (DB baseline) up to 2 years 2 months in the DB phase
  Change from DB baseline in SF measured by CSFQ-14 total score and SF domain scores over time will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (95):
- United States (31):
  - Preferred Research Partners, Little Rock, Arkansas
  - Wake Research PRI Encino, Encino, California
  - Wr Pri Llc, Newport Beach, California
  - ATP Clinical Research, Orange, California
  - Myndful Research, Redlands, California
  - Artemis Institute for Clinical Research, San Diego, California
  - UHC Research, Doral, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - GTL Medical and Research Group, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Harmony Clinical Research Inc, North Miami Beach, Florida
  - APG Research LLC, Orlando, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Synexus Clinical Research US Inc, Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Psychiatric Medicine Associates LLC, Skokie, Illinois
  - Continental Clinical Solutions, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Missouri Health Care, Columbia, Missouri
  - IMA Clinical Research PC, Albuquerque, New Mexico
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - Insight Clinical Trials, Independence, Ohio
  - Laureate Institute for Brain Research, Tulsa, Oklahoma
  - Keystone Clinical Studies LLC, Plymouth Meeting, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - InSite Clinical Research LLC, DeSoto, Texas
  - Earle Research, Friendswood, Texas
  - Alpine Research Organization, Clinton, Utah
  - Elligo Integrated Research Sites Integrated Clinical Research LLC Integrated Psych, St. George, Utah
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Centro Medico Instituto Modelo de Neurologia y Neurorehabilitacion, Córdoba
- Belgium (5):
  - Anima, Alken
  - AZ Sint-Lucas, Assebroek
  - UZ Brussel, Brussels
  - AZ Oudenaarde, Oudenaarde
  - Vitaz, Sint-Niklaas
- Brazil (2):
  - CAEP Centro Avancado De Estudos E Pesquisas, Campinas
  - Centro Integrado Facili, São Bernardo do Campo
- Bulgaria (5):
  - Mental Health Center - Rousse, Rousse
  - Medical Centre Akademika EOOD, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Diagnostic Consulting Center Mladost - M Varna, Varna
  - Mental Health Center - Vratsa EOOD, Vratsa
- France (5):
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Hopital la Colombiere, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - CHS du Rouvray, Sotteville-lès-Rouen
  - Hopital Sainte Musse, Toulon
- Germany (9):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Praxis Dr. med. Kirsten Hahn, Berlin
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Chemnitz
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Klinische Forschung Hamburg, Hamburg
  - Oberhavel Kliniken GmbH, Hennigsdorf
  - Universitaetsklinikum Muenster, Münster
  - Boehm Peters Praxis fur Psychiatrie Psychotherapie Neurologie PartGmbB, Rosenheim
  - Klinische Forschung Schwerin GmbH, Schwerin
- Greece (5):
  - Eginitio Hospital, Athens
  - Attikon University General Hospital of Attica, Athens
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - G Papanikolaou Hospital of Thessaloniki, Thessaloniki
- Mexico (4):
  - Hospital Aranda de la Parra S A de C V, León
  - Ketamine Mexico S de RL de C V, Mexico City
  - Human Science Research Trials S de RL de CV, México
  - cit NEUROPSIQUE, Monterrey
- Poland (10):
  - Osrodek Badan Klinicznych CLINSANTE S C Ewa Galczak Nowak Malgorzata Trzaska, Bydgoszcz
  - NZOZ Euromedica Grudziadz, Grudziądz
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Centrum Medyczne Luxmed Sp z o o, Lublin
  - Praktyka Lekarska dr n med Malgorzata Wojtanowska Bogacka, Poznan
  - Indywidualna Specjalistyczna Praktyka Lekarska Agnieszka Remlinger Molenda, Suchy Las
  - Care Access Warszawa, Warsaw
  - Szpital Nowowiejski Osrodek Badan Klinicznych, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Centrum Zdrowia Mosty, Wroclaw
- Romania (7):
  - Spitalul Clinic de Psihiatrie Prof Dr Alexandru Obregia, Bucharest
  - Centrul de Evaluarea si Tratament al Toxicodependentelor pentru Tineri Sf. Stelian, Bucharest
  - Centrul Medical Melchisedec, Craiova
  - Spitalul Clinic de Neuropsihiatrie, Craiova
  - CMI Dr. Sarpe Marcel-Claudiu, Focşani
  - Spitalul De Psihiatrie Elisabeta Doamna Galaţi, Galați
  - Spitalul Clinic De Psihiatrie Doctor Gheorghe Preda, Sibiu
- Spain (9):
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. Univ. La Paz, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Son Espases, Palma
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. El Bierzo, Ponferrada
  - Hosp. Royo Villanova, Zaragoza
- Erenkoy Mental Health Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency